# STUDY TITLE: A MULTI-CENTER, PROSPECTIVE STUDY TO EVALUATE THE SAFETY AND EFFECTIVENESS OF MULTI -TREATMENT REGIMEN WITH ZELTIQ AESTHETICS, INC. RAPID ACOUSTIC PULSE (RAP)™ DEVICE FOR THE IMPROVEMENT IN THE APPEARANCE OF CELLULITE

PROTOCOL NUMBER: 2022-01

Rev: 02

DATE: March 20, 2024 Contact:

Sponsor: ZELTIQ Aesthetics, Inc. 4410 Rosewood Drive Pleasanton, CA 94588

## CONFIDENTIALITY STATEMENT

This document contains confidential information that is the property of ZELTIQ Aesthetics, Inc., and may not be disclosed to anyone other than the recipient clinical Investigator or his or her staff.

This information cannot be used for any purpose other than the evaluation and conduct of the clinical investigation without the prior written consent of ZELTIQ Aesthetics, Inc.

# TABLE OF CONTENTS

| INVESTIGATOR'S STATEMENT OF AGREEMENT | 5 |
|---|---|
| CLINICAL SITES | 6 |
| STUDY SYNOPSIS | 7 |
| INTRODUCTION OVERVIEW | 11 |
| CELLULITE | |
| ZELTIQ AESTHETICS, INC.'S RAPID ACOUSTIC PULSE (RAP) DEVICE WITH CEL | LULITE |
| CARTRIDGE | |
| PHYSICAL EFFECTSPROOF OF CONCEPT (POC) OF SAFETY AND TOLERABILITY OF RAP CELLULITE | |
| CLINICAL TRIAL | |
| SAFETY CONCLUSION | |
| PIVOTAL STUDY OF SAFETY AND EFFICACY OF RAP CELLULITE CLINICAL TRIA | L13 |
| STUDY DESIGN | 17 |
| SELECTION OF STUDY POPULATION | 17 |
| INCLUSION CRITERIA | |
| EXCLUSION CRITERIA | |
| STUDY VISITSVISIT 1 BASELINE SCREENING AND CONSENT FORM (DAY -30 TO DAY 0) | |
| VISIT 2 TREATMENT | |
| VISIT 3 FOLLOW UP VISIT 4-WEEKS POST 1ST TREATMENT (+/- 14 DAYS) AND 2 <sup>N</sup> | D |
| TREATMENT | |
| VISIT 4 FOLLOW UP VISIT 12-WEEKS POST 2 <sup>ND</sup> TREATMENT (+/- 14 DAYS) | |
| VISIT 6 FOLLOW UP VISIT 52-WEEKS POST 2 <sup>ND</sup> TREATMENT (+/- 14 DAYS) | |
| RISKS AND BENEFITS | |
| KNOWN SIDE EFFECTS OF RAP TREATMENTERROR! BOOKMARK NO KNOWN TREATMENT ADVERSE EVENTSERROR! BOOKMARK NO | |
| RISK MITIGATIONSERROR. | |
| REPORTING ADVERSE EVENTS AND COMPLICATIONS | |
| ADVERSE EVENTS | |
| DEVICE MALFUNCTIONS | 27 |
| STUDY PARTICIPANT INFORMED CONSENT | 27 |
| RECORDS MANAGEMENT | 28 |
| INVESTIGATIONAL DEVICE ACCOUNTABILITY AND STORAGE | |
| REGULATORY AND ETHICAL COMPLIANCE | |
| QUALITY ASSURANCE AND MONITORING | |
| STUDY RESULTS/ANALYSIS | |
| SUSPENSION OR PREMATURE TERMINATION OF STUDY | |
| PUBLICATION POLICY | |
| STUDY COMPLETION | |
| REFERENCES | |
| TABLES | |
| TIMELINE AND EVENTS SCHEDULE | |
| STUDY SCALES AND ASSESSMENTS | 33 |

#### INVESTIGATOR'S STATEMENT OF AGREEMENT

I have read the foregoing protocol and agree that it contains all necessary details for conducting the study. I will conduct the study as outlined herein and will complete the study within the time designated.

I agree to conduct this protocol in accordance with local regulations, external standards and applicable ICH and Good Clinical Practice (GCP) guidelines.

I will provide copies of the protocol, including any amendments, and all pertinent information to all individuals responsible to me who assist in the conduct of this study. I will discuss this material with them to ensure they are fully informed regarding the ZELTIQ Aesthetics, Inc. device and the conduct of the study.

I further agree to provide access to ZELTIQ Aesthetics Inc, its designees, or regulatory authorities to any source documents from which case report form information may have been generated.

I agree to maintain the confidentiality of all information received or developed in connection with this protocol.

| Date | |
|------|------|
| | Date |

# **CLINICAL SITES**



# STUDY SYNOPSIS

| Purpose Primary | The purpose of this multi-site clinical study is to evaluate the safety and effectiveness in the appearance of cellulite. |
|---|---|
| Effectiveness Objective | The primary effectiveness objective will demonstrate improvement in the appearance of cellulite as determined by correct identification of baseline vs 12-weeks post final treatment images. |
| Secondary<br>Objectives | Evaluate the safety of the RAP device for cellulite treatments The secondary effectiveness objective: will demonstrate improvement in the appearance of cellulite as determined by the study participants completing the Participant Satisfaction Survey |
| | photos of the thighs and/or buttocks area will serve as a control. |
| Study Design | Non-significant risk, multi-site, prospective clinical trial. |
| Planned Number<br>of Sites /<br>Countries | Four (4) clinical trial sites located in the United States. |
| Planned Number<br>of Participants/<br>Treatment Areas | Up to sixty (60) participant |















# PROTOCOL 2022-01 STUDY OBJECTIVES AND ENDPOINTS

| Primary Objective | Primary Outcome Endpoint |
|---|---|
| RAP treatment effectiveness: The primary effectiveness objective will demonstrate improvement in the appearance of cellulite as determined by correct identification of baseline vs 12-weeks post final treatment images | |







#### STUDY DESIGN

This is a non-significant risk, multi-center, multi-treatment (2 treatment sessions) prospective trial for safety, and effectiveness using ZELTIQ Aesthetics, Inc.'s RAP device for the improvement in the appearance of cellulite performed at up to four (4) clinical research sites in the United States.

Up to sixty (60) healthy participants will be enrolled in this study.

Participants who sign the informed consent form and meet all the eligibility criteria will be enrolled in the study.

# **Selection of Study Population**

The clinical study can fulfill its objectives only if appropriate participants are enrolled.

The following criteria are designed to select participants for whom protocol requirements are considered appropriate.

Participants who meet all inclusion criteria and none of the exclusion criteria will be enrolled in the study and assigned a participant No./ID in sequential order (i.e., 01, 02, 03, etc.)

#### **Inclusion Criteria**

- Healthy candidates
- Seeking treatment of cellulite in the thigh and/or buttock areas



• Participant must be able to provide written informed consent, understand and comply with all study-related procedures and follow-up visits.

# **Exclusion Criteria**



 Any other condition/disease/situation which, as deemed by the PI, would preclude participant from safely participating in or completing the study visits or that may confound study results.









# UNSCHEDULED VISITS

An unscheduled visit may be performed at any time during the study at the participant's request or as deemed necessary by the study investigator. The date and reason for the visit will be recorded in the source document.

#### PARTICIPANT WITHDRAWL AND EARLY TERMINATION

Participants may withdraw from the study at any time at their own request or withdrawn from at any time at the discretion of the Investigator for safety, behavioral, or administrative reasons. The Investigator should inquire about reason for withdrawal, request the participant to return for a final visit, and follow up with any unresolved adverse events. The Investigator should notify the Sponsor of any participants withdrawal or discontinuance.









#### **Adverse Events**

The Investigator is responsible for the detection and documentation of events meeting the criteria and definition of an AE or SAE, as provided in this protocol. During the study when there is a safety evaluation, the Investigator or site staff will be responsible for detecting, documenting, and reporting AEs and SAEs as detailed in this Section of the protocol.

At the treatment and follow-up visits, participants will be assessed for known physiological responses and adverse events.

## Adverse Event (AE)

- An adverse event (AE) is defined as any unfavorable or unintended sign, symptom, or disease that occurs or is reported by the participant to have occurred, or a worsening of a pre-existing condition. An adverse event may or may not be related to the study treatment.
- AEs will be elicited through direct questioning and participant reports. Any abnormality in physical examination findings that the investigator believes is clinically significant (CS) to the research participant and that occurred after initiation of the first study treatment will be reported as AEs. Abnormal findings that are NOT clinically significant should not be recorded as an AE.

#### Adverse Device Effect (ADE)

O An ADE is defined as an adverse event related to the use of an investigational medical device. This definition includes any adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device as well as any event resulting from use error or from intentional misuse of the investigational medical device. This includes "comparator" if the comparator is a medical device.

#### 1. Reporting of Adverse Events

- Report initiation for all AEs and SAEs will begin at the time of the first treatment and continue until the end of the final study observation visit. All events will be followed to resolution or until the participant completes the study. A final assessment of outcome will be made at that time.
- O All AEs must be recorded in the participant's medical records and in the case report form. AEs will be reported using customary medical terminology along with the following information: the onset and end dates, whether the event is considered to be a SAE, the impact the event had on study treatment, the

severity of the event, the causality of the event, whether treatment was given as a result of the event, and the outcome of the event.

### 2. Impact on Study Treatment

The impact the event had on the study treatment will be assessed as either: none, study treatment interrupted, study treatment discontinued, or not applicable.
 The "not applicable" assessment will be used only when the participant is in the observation phase of the protocol.

#### 3. Causality Assessment

- AEs will be assigned a relationship (causality) to the study treatment. The Investigator will be responsible for determining the relationship between an AE and the study treatment. The type of event, organ system affected, and timing of onset of the event will be factors in assessing the likelihood that an AE is related to the study treatment. Relationship of AEs to study treatment will be classified as follows:
  - i. Definitely related: This category applies to those AEs that the Investigator feels are incontrovertibly related to the study treatment. An AE may be assigned an attribution of definitely related if or when it meets all of the following criteria: (1) it follows a reasonable temporal sequence from administration of the study treatment; (2) it could not be reasonably explained by the known characteristics of the participant's clinical state, environmental or toxic factors, or other modes of therapy administered to the participant; (3) it follows a known response pattern to treatment with the study treatment.
  - ii. Probably related: This category applies to those AEs which, after careful medical consideration at the time they are evaluated, are felt with a high degree of certainty to be related to the study treatment. An AE may be considered probable if or when (must have three): (1) it follows a reasonable temporal sequence from administration of the study treatment. (2) It could not readily have been produced by participant's clinical state, environmental or toxic factors, or other therapies administered to the participant. (3) Disappears or is decreased upon discontinuation of the study treatment. (4) It follows a known response pattern to treatment with the study treatment.
  - iii. Possibly related: This category applies to those AEs which, after careful medical consideration at the time they are evaluated, are judged unlikely but cannot be ruled out with certainty to the study treatment. An AE may be considered possible if or when (must have two): (1) it follows a reasonable temporal sequence from administration of the study treatment. (2) It could not readily have been produced by participant's clinical state, environmental or toxic factors, or other therapies administered to the participant. (3) Disappears or is decreased upon discontinuation of the study treatment. (4) It follows a known response pattern to treatment with the study treatment.

- iv. Remotely related: In general, this category can be considered applicable to those AEs which, after careful medical consideration at the time they are evaluated, are judged likely to be unrelated to the study treatment. An AE may be considered unlikely if or when (must have two): (1) it does not follow a reasonable temporal sequence from administration of the study treatment. (2) It could not readily have been produced by participant's clinical state, environmental or toxic factors, or other therapies administered to the participant. (3) Disappears or is decreased upon discontinuation of the study treatment. (4) It does not follow a known response pattern to treatment with the study treatment.
- v. Unrelated: This category applies to those AEs which, after careful consideration at the time they are evaluated, are clearly and incontrovertibly due to extraneous causes (disease, environment, etc.) and determined with certainty to have no relationship to the study treatment.

#### 4. Outcome Assessment

The outcome of the event will be assessed as either: resolved, resolved with sequelae, ongoing, or death. Only one AE per participant is allowed to have an outcome assessment as "death." If there are multiple causes of death for a given participant, only the primary cause of death will have an outcome of death.

#### 5. Serious Adverse Events

- o A Serious Adverse Event (SAE) is defined as any AE that:
  - i. Results in death
  - ii. Is life threatening (the participant is at immediate risk of dying from the adverse experience)
  - iii. Requires participant hospitalization or prolongs existing hospitalization
  - iv. Results in persistent or significant disability/incapacity
  - v. Is a congenital anomaly/birth defect
  - vi. Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function

#### 6. Reporting SAEs

- The Investigator is required to report all SAEs that occur from RAP treatment through 30 days post end of study. Once the investigator becomes aware of an SAE, he/she must report the SAE to the Sponsor, ZELTIQ Aesthetics, Inc. within 24 hours.
  - Contact Information:
    - Email:
    - Phone:

- o The Sponsor ZELTIQ Aesthetics, Inc. may request additional supporting documentation as it becomes available, such as lab reports, electrocardiogram reports, discharge summary, hospital notes, etc., if applicable. Additional followup information as it becomes available must be reported to the same phone number and contact info listed at the beginning of this document.
- The Investigator is also responsible for reporting all SAEs to the appropriate Institutional Review Board (IRB) in accordance with local laws and regulations. The Investigator is responsible for maintaining documentation in the study file that indicates the IRB has been properly notified.

#### 7. SAE Follow-up

- O All participants experiencing an SAE, including discontinued participants, must be closely followed until sufficient information is obtained to indicate a return to normal status or until the event stabilizes at a level acceptable to the investigator, i.e., recovery, return to baseline status, no further improvement expected, or death.
- For each SAE indicated as an unresolved event on the initial report, regardless of
  whether the participant completed the study or withdrew, the site should submit
  a follow-up report with updated information.



#### STUDY PARTICIPANT INFORMED CONSENT

All eligible participants must sign the informed consent form prior to enrollment in the study. The participant and the Investigator or designee will discuss the benefits and risks of the study and review the participant consent form to ensure the participant understands the scope of the study. It is the Investigator's or designee's responsibility to ensure that participants understand that participation in the study is voluntary, and that the quality of their medical care will not be adversely affected if they decline to participate in the study. Adequate time for any questions and explanations will be provided. Participants will have the opportunity to discuss the study with their surrogates and have time to think about it prior to participating. Participants may withdraw their consent at any time throughout the course of treatment. Once the participant understands the informed consent, he/she will be allowed to voluntarily agree to participate by signing the document. The investigator/designee is responsible for obtaining informed consent prior to enrollment in the study and ensuring that the participant has a copy of the document for their records. The participant is considered enrolled in the study after the informed consent has been signed and it has been verified that the participant meets all inclusion criteria and none of the exclusion criteria.

#### RECORDS MANAGEMENT

**Study Records Retention**: Each site will maintain appropriate medical records for this study in accordance with institutional requirements including, but not limited to, hospital records, laboratory tests, pharmacy dispensing records, x-rays, and clinical charts. As part of study participation, each site will permit the Sponsor ZELTIQ Aesthetics, Inc., or its designee, to examine (and when required by applicable law, to copy) clinical records for the purposes of quality assurance reviews, audits and evaluation of study safety and progress.

- i. Essential documents, as listed below, must be retained by the site until at least 2 years after completion or termination of the investigation, or longer if:
- ii. Advised by the Sponsor or designee. If the Investigator relocates, retires, or for any reason cannot keep study records, the records may be transferred to an acceptable designee. The Sponsor or its designee must be notified in writing of the name, address, and telephone number of the person designated to retain the study records. By signing the protocol, the Investigator agrees to adhere to the document retention procedures.
- iii. Essential documents may include:
  - 1. IRB approvals for the study protocol and all amendments
  - 2. Participant's informed consent forms
  - 3. All source documents
  - 4. Case Report Forms
  - 5. Data change forms or data queries
  - 6. Monitoring logs and appointment schedules
  - 7. Investigators CVs, medical license information, and financial disclosure documentation
  - 8. All sponsor representative/investigator correspondence, including telephone logs
  - 9. Any other pertinent study documents

**Protocol Deviations**: Protocol deviations occur when there are variations in the approved study protocol, criteria, or procedure. An example of this would be a participant visit conducted outside the follow-up schedule. As protocol deviations may increase the risk or decrease the benefit of the intervention and/or affect the participant's rights, safety, welfare and/or integrity of the resultant data, investigators are required to record and report all incidences in a deviation log for adjudication during data analysis.

iv. All protocol deviations must be reported to Sponsor in a timely manner of their occurrence. Evaluation of the deviation and its impact on the study protocol will be adjudicated on a case-by-case basis. Data discrepancies or questions resulting from reported protocol deviations will be managed between Sponsor and the site investigator or their designee.

#### INVESTIGATIONAL DEVICE ACCOUNTABILITY AND STORAGE

The Sponsor will maintain full device accountability. The Investigator will maintain adequate records documenting all materials received and returned, and shipping information of the device. All used materials will be discarded by the Investigator after each treatment has been completed.

## REGULATORY AND ETHICAL COMPLIANCE

- 1. The Study will comply with all instructions, regulations, and agreements in this protocol. In addition, the study will comply with all local regulations, external standards and applicable ICH and Good Clinical Practice (GCP) guidelines.
- Institutional Review Board: The site that is participating in this study must have this
  protocol and the associated informed consent approved through the IRB. Any
  amendments to the protocol or informed consent will be routed through IRB for
  approval prior to use.
- 3. Participant Confidentiality: Participant confidentiality for all data collected during the course of treatment will be maintained by the Investigator, on-site staff, and the Sponsor. All pictures of the participant's test areas will be de-identified, secure, privileged, and compliant with all HIPAA guidelines. A unique participant identification (ID) code will be assigned to each participant in the study. This ID code will be used throughout the course of treatment to ensure that no identifying information exists on any Case Report Forms. The document which contains the participant ID key will be stored in a locked cabinet and will only be accessible by authorized study personnel. Private and confidential information about each participant will be preserved in any report or publication of the clinical investigation data.
- 4. <u>Investigator Conflict of Interest:</u> The proposed study will be conducted in accordance with signed investigator statements.
- 5. Funding Source: Funding for this study is provided by ZELTIQ Aesthetics, Inc.
- 6. <u>Changes to Final Protocol:</u> ZELTIQ Aesthetics, Inc. may amend the protocol at any time. All protocol modifications that could potentially affect data collection practices, study scope, participant safety, or scientific quality will be submitted to the IRB for approval prior to implementing the changes.







#### SUSPENSION OR PREMATURE TERMINATION OF STUDY

The Sponsor reserves the right to suspend or prematurely terminate the study in its entirely or at an investigational site for significant and documented reasons. An Investigator, IRB, or regulatory authority may suspend or prematurely terminate participation in the clinical investigation for which they are responsible at any time in collaboration with the Sponsor.



## STUDY COMPLETION

The IRB must be notified of completion of this study.

























